CLINICAL TRIAL: NCT02080078
Title: A Phase I, Single-center, Non-randomized, Open-label Study to Determine the Lowest Effective Theophylline Dose That Decreased Erlotinib's Diarrhea at the Standard Dose of 150 mg/Day and to Determine the Highest Erlotinib Dose in Combination With Theophylline That Can be Administered to Patients
Brief Title: A Phase I Dose Escalation Study of Erlotinib in Combination With Theophylline
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: REB decision
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Theophylline 1.0
Record Dates: First submitted 2014-02-12; First posted 2014-03-06 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Non-small Cell Lung Cancer; Advanced Solid Malignancies
Keywords: Erlotinib; Theophylline; Diarrhea
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Diarrhea | interventions — Theophylline; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Increasing dose of Theophylline (Experimental): Patients will be put on the standard dose of 150 mg/day of erlotinib. Patients will be entered into the study on different dose levels of theophylline (100 mg/bid, 150 mg/bid, 200 mg/bid, or 200 mg/tid) for 28 days to find what is the lowest dose that effectively controls the diarrhea caused by erlotinib.
  Interventions: Drug: Theophylline; Drug: Erlotinib
- Increasing dose of erlotinib (Experimental): Patients will be kept on a specified dose of theophylline while the dose of erlotinib increases in each group of patients enrolled (200 mg/qd, 225 mg/qd, or 250 mg/qd) for 28 days to determine what the maximum dose of erlotinib that can be given with theophylline and maintain a safety profile.
  Interventions: Drug: Theophylline; Drug: Erlotinib

INTERVENTIONS:
Drug: Theophylline
  Other Names: Theo-Dur
Drug: Erlotinib
  Other Names: Tarceva

SUMMARY:
This study is to determine the use of theophylline in patients with NSCLC and advanced solid malignancies and whether treatment with theophylline will help lower or diminish the side effect of diarrhea in patients taking erlotinib. Patients will be enrolled in one of two parts of the study to verify the lowest dose of theophylline that is effective and the highest dose of erlotinib that can be tolerated with theophylline. If this study shows that theophylline is able to inhibit erlotinib induced diarrhea, it will help demonstrate that patients using the tyrosine kinase inhibitor (TKIs), erlotinib, can use it effectively at higher doses without experiencing severe diarrhea.

DETAILED DESCRIPTION:
Erlotinib is a tyrosine kinase inhibitor (TKI), which is a newer, effective treatment for cancer patients. TKIs are the only class of anticancer drugs that are predominately used as single agents. TKIs were hoped to lack side effects but can cause severe enough diarrhea that patients frequently stop treatment, even if TKIs are controlling their cancer. TKIs inhibit nucleoside transporters (NTs), perturbing regulation of adenosine levels in the intestine. It is possible that the reason for the inability to use TKIs in combination therapies has been their additive effects on NTs causing unacceptable diarrhea. It has been shown that TKIs are potent NT inhibitors, therefore it will theoretically inhibit NTs of intestinal epithelial cells causing an accumulation of extracellular adenosine resulting in chloride secretory diarrhea. If this hypothesis is correct, it has profound implications for oncology, since diarrhea is one of the dose-limiting toxicities of TKIs. It has been shown that co-incubating cells with 8-phenyltheophylline (8PT), which is an A2B adenosine receptor antagonist, block chloride secretion caused by nitrobenzyl-mercaptopurine ribonucleoside (NBMPR). Theophylline is also a methylxanthine and is a commercially available and licensed example of a 8PT. As it is already known that erlotinib is effective, it is used as a control factor in the first arm of the study and will be increased in the second arm to see what the maximally tolerated dose is when in combination with a controlled dose of theophylline.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any study specific procedure. Patients must be able to understand and willing to sign the written informed consent.
* Subjects with histologically confirmed, advanced, metastatic or refractory solid malignancy who are not candidates for standard therapy or patients with advanced or recurrent NSCLC
* Male / female subject ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2.
* Women of childbearing potential and men must agree to use adequate contraception since signing of the informed consent form until at least 8 weeks after the last study drug administration. The investigator or a designated associate is requested to advise the subject how to achieve an adequate birth control. Adequate contraception is defined in the study as any medically recommended method (or combination of methods) as per standard of care.
* Women of childbearing potential must have a negative urine pregnancy test performed within 7 days before start of study treatment.
* Life expectancy at least 8 weeks
* Adequate bone marrow, renal function and liver function as assessed by the following laboratory requirements conducted within 7 days of starting the study treatment:
* Platelet count ≥ 100.000/cubic millimeters (mm3), hemoglobin (Hb) ≥ 9.0 g/dl, absolute neutrophil count (ANC) ≥ 1500/mm3.
* Total bilirubin ≤ 1.5 x the upper limit of normal range (ULN). Mildly elevated total bilirubin (<6 mg/dL) is allowed if Gilbert's syndrome is documented.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤5 x ULN for subjects whose cancer involves their liver including liver metastasis)
* Alkaline phosphatase limit ≤ 2.5 x ULN (≤ 5 x ULN for subjects whose cancer involves their liver including liver metastasis).
* Estimated glomerular filtration rate (eGFR) ≥ 50 mL/min as calculated using the Cockcroft-Gault formula
* International normalized ratio (INR) ≤ 1.5 x ULN. Subjects who are being treated with heparin are allowed to participate.

Exclusion Criteria:

* Prior treatment with erlotinib. Patients permanently withdrawn from study participation will not be allowed to re-enter the study.
* Symptomatic metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, has no evidence of tumor growth on an imaging study within 4 weeks prior to study entry and is not on dexamethasone and clinically stable with respect to the tumor at the time of study entry.
* Major surgery, open biopsy, or significant traumatic injury within 28 days before starting the study treatment
* History of organ allograft
* Non-healing wound, skin ulcer, or bone fracture
* Uncontrolled concurrent medical illness including uncontrolled hypertension defined as systolic blood pressure >150 millimeter of mercury (mmHg) or diastolic blood pressure >90 mmHg, despite medical management
* History of cardiac disease: congestive heart failure > NYHA (New York Heart Association) Class II; unstable angina (symptoms of angina at rest), new-onset angina (within the last 3 months), myocardial infarction within the past 6 months prior to screening (Visit 1); cardiac ventricular arrhythmias requiring anti-arrhythmic therapy (except for beta-blockers and digoxin)
* Pleural effusion or ascites that causes respiratory compromise (NCI-CTCAE version 4.0 Grade ≥ 2 dyspnea)
* Interstitial lung disease with ongoing signs and symptoms within 28 days before starting the study treatment
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before the start of study medication
* Subjects with evidence or history of bleeding diathesis; any hemorrhage or bleeding event CTCAE Grade ≥ 3 or higher within 4 weeks of start of investigational treatment
* Dehydration CTCAE Grade ≥ 1
* Unresolved toxicity higher than NCI-CTCAE version 4.0 Grade 1 (excluding alopecia, anemia or lymphopenia) attributed to any prior systemic or radiation therapy or other medical or surgical procedure
* Known hypersensitivity to erlotinib, study drug class, or excipients in the formulation
* Ongoing or active infection (bacterial, fungal, or viral, e.g. human immunodeficiency virus (HIV)) of NCI-CTCAE version 4.0 Grade ≥ 2
* Seizure disorder requiring anticonvulsant therapy (such as steroids or anti-epileptics)
* Pregnancy and lactation (breast feeding)
* During the study, no other anticancer treatment, including any investigational new drugs, is allowed. Anticancer therapy is defined as any agent or combination of agents with clinically proven anticancer activity. Systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and hormonal therapy during this trial or within 28 days or 5 drug half-lives (if drug half-life in subjects is known), whichever is shorter (or within 6 weeks for mitomycin C) before start of the study treatment.
* Use of hematopoietic growth factors, such as G-CSF (granulocyte colony-stimulating factor), GM-CSF (granulocyte-macrophage colony-stimulating factor), erythropoietin, and interleukin (Il-2, IL-3), within 3 weeks prior to first dose. G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator; however, they may not be substituted for a required dose reduction. Subjects taking chronic erythropoietin consistent with institutional guidelines can be included.
* Close affiliation with the investigational site; e.g. a close relative of the investigator or a dependent person (e.g. employee or student of the investigational site)
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Inability to swallow oral medications
* Inflammatory bowel disease or other disorders associated with chronic diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09; Primary Completion 2019-03-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
The lowest effective dose of theophylline that will prevent or maximally ameliorate erlotinib's diarrhea at the standard dose of erlotinib at 150 mg/day taken daily for 28 days every 28 days | 28 days

SECONDARY OUTCOMES:
The highest dose of erlotinib that can be administered with theophylline and can be administered with an acceptable safety profile | 28 days
  Once the lowest effective dose of theophylline that will prevent or maximally ameliorate erlotinib's diarrhea at 150 mg/day taken daily for 28 days is determined, we will determine what is the highest dose of erlotinib that can be administered with theophylline that can be administered with an acceptable safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sawyer, MD, Principal Investigator — Alberta Health services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada